CLINICAL TRIAL: NCT01356667
Title: Drum-Assisted Recovery Therapy for Native Americans
Brief Title: Drum-Assisted Therapy for Native Americans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study period is over and recruitment was stopped due to time constraints.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Dickerson, Assistant Research Psychiatrist, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DARTNA
Record Dates: First submitted 2011-04-26; First posted 2011-05-19 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-05

CONDITIONS: Substance Use Disorders
Keywords: American Indians; Native Americans; substance abuse; culture
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment-As-Usual (Active Comparator): Substance Abuse treatment typically received
  Interventions: Behavioral: Treatment-As-Usual
- DARTNA (Experimental): 12-week DARTNA program
  Interventions: Behavioral: DARTNA

INTERVENTIONS:
Behavioral: DARTNA — 3-hour protocol provided 2x/week over 12 weeks
  Arms: DARTNA
Behavioral: Treatment-As-Usual — Participants will receive typical substance abuse behavior treatment interventions typically provided to patients including individual counseling, group therapy, and standard culturally-based interventions.
  Arms: Treatment-As-Usual

SUMMARY:
Drum-Assisted Recovery Therapy for Native Americans (DARTNA) is an R-21 NIH/NCCAM-funded study aimed to complete the development and pilot a new substance abuse treatment protocol utilizing drumming for American Indians/Alaska Natives with substance use disorders. The study includes activities to complete the protocol, followed by a randomized-controlled clinical trial.

DETAILED DESCRIPTION:
During year 1, this study consists of a series of focus groups conducted among American Indians/Alaska Natives with substance use disorders, providers serving AI/ANs with substance use disorders, and a Community Advisory Board. These focus groups are conducted in order to obtain feedback with regard to the initial DARTNA treatment protocol. These focus groups are then followed by a pretest of DARTNA among 10 AI/ANs with substance use disorders followed by a series of focus groups to finalize the development of DARTNA. During year 2, a randomized controlled will be conducted among 30 AI/ANs receiving the DARTNA treatment protocol vs. 30 AI/ANs receiving treatment-as-usual at United American Indian Involvement, Inc. in Los Angeles.

ELIGIBILITY:
Inclusion Criteria:

* meeting Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR; American Psychiatric Association, 2000) criteria of current alcohol or drug abuse or dependence
* self-identifying as at least ¼ American Indian/Alaska Native heritage
* seeking treatment for alcohol or drug abuse
* being at least 18 years old. Clients will be assessed for suitability for outpatient treatment.

Exclusion Criteria:

* have a psychiatric conditions that is not suitable for outpatient treatment (e.g., if they require inpatient rehabilitation treatment, have significant psychiatric disorders, require medical detoxification, or have significant medical problems)
* have a current suicidal ideation/plan as assessed by the ASI or BSI
* are mandated by the court to obtain treatment for substance abuse where such mandate requires the results of urine toxicology tests to be reported to the court
* expectation that the participant will fail to complete the study protocol due to probable incarceration or relocation from the clinic area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Dickerson, D.O., M.P.H., Principal Investigator — University of California, Los Angeles
Locations (1):
- United American Indian Involvement, Inc., Los Angeles, California, United States

REFERENCES:
- [Derived] Dickerson DL, D'Amico EJ, Klein DJ, Johnson CL, Hale B, Ye F. Mental Health, Physical Health, and Cultural Characteristics Among American Indians/Alaska Natives Seeking Substance Use Treatment in an Urban Setting: A Descriptive Study. Community Ment Health J. 2021 Jul;57(5):937-947. doi: 10.1007/s10597-020-00688-3. Epub 2020 Jul 27. PMID 32720004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted from Sept, 2011-August 2012 and took place at United American Indian Involvement, Inc.
Pre-assignment Details: No enrolled participants were excluded from the trial before assignment to groups.
Groups:
- Treatment-As-Usual: Substance Abuse treatment typically received at United American Indian Involvement (UAII)
- Drum-Assisted Recovery Therapy for Native Americans: 12-week treatment protocol consisting of drum therapy for Native Americans
Period: Overall Study
Arm/Group | Treatment-As-Usual | Drum-Assisted Recovery Therapy for Native Americans
Started | 4 | 6
Completed | 0 | 0
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-As-Usual | Drum-Assisted Recovery Therapy for Native Americans | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (9.0) | 50.3 (3.9) | 44.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Drug and Alcohol Use as a Measure of Treatment Effectiveness
Description: Urine drug screens and breathalyzers will be obtained from patients in order to determine their recent drug and alcohol use.
Time Frame: Change from Baseline in Drug and Alcohol use at 6 months
Population: Please be advised that this clincial trial was terminated prior to finalization of any research procedures.
Arm/Group | Treatment-As-Usual | Drum-Assisted Recovery Therapy for Native Americans
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Knowledge of Alcoholics Anonymous Concepts as a Measure of Protocol Comprehension
Description: The General Alcoholics Anonymous Tools of Recovery (GAATOR 2.1) will be provided in order to determine and track patient's knowledge of the 12-steps during their participation in the DARTNA treatment program.
Time Frame: Change from Baseline in Knowledge of Alcoholics Anonymous at 12 weeks
Population: Please be advised that this clincial trial was terminated prior to finalization of any research procedures.
Arm/Group | Treatment-As-Usual | Drum-Assisted Recovery Therapy for Native Americans
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mental Health and Psychosocial Characteristics as Measured by the Addiction Severity Index, Native American Version and Brief Symptom Inventory.
Description: The Addiction Severity Index, Native American Version will be utilized to assess problem severity in alcohol use, drug use, employment, family and social relationships, legal, psychological, and medical status. In addition, additional information with regards to mental health characteristics will be obtained from the Brief Symptom Inventory.
Time Frame: Change from Baseline in Mental Health and psychosocial characteristics at 6 months
Population: Please be advised that this clincial trial was terminated prior to finalization of any research procedures.
Arm/Group | Treatment-As-Usual | DARTNA
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment-As-Usual | Drum-Assisted Recovery Therapy for Native Americans
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/4 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes